CLINICAL TRIAL: NCT06408649
Title: Post-market Clinical Follow-up Study of Alcon TOTAL30® Spherical Contact Lenses (Lehfilcon A) and TOTAL30® for Astigmatism Contact Lenses (Lehfilcon A)
Brief Title: Post-market Clinical Follow-up Study of Alcon TOTAL30® Contact Lenses (Lehfilcon A)
Status: Terminated | Type: Observational
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLY935-N001
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Ametropia; Myopia; Hyperopia; Astigmatism
Keywords: Contact lenses
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TOTAL30 Sphere: Lehfilcon A spherical contact lenses worn in both eyes in a real-world setting
  Interventions: Device: Lehfilcon A spherical contact lenses
- TOTAL30 for Astigmatism: Lehfilcon A toric contact lenses worn in both eyes in a real-world setting
  Interventions: Device: Lehfilcon A toric contact lenses

INTERVENTIONS:
Device: Lehfilcon A spherical contact lenses — Silicone hydrogel contact lenses for the correction of ametropia (myopia or hyperopia)
  Other Names: TOTAL30® Spherical Contact Lenses
  Groups: TOTAL30 Sphere
Device: Lehfilcon A toric contact lenses — Silicone hydrogel contact lenses for the correction of ametropia (myopia or hyperopia) with astigmatism
  Other Names: TOTAL30® for Astigmatism Contact Lenses
  Groups: TOTAL30 for Astigmatism

SUMMARY:
The purpose of this Post-Market Clinical Follow-Up (PMCF) study is to continuously assess the visual performance and safety of TOTAL30 Sphere and TOTAL30 for Astigmatism contact lenses in a real-world setting across a broad variety of patients through routine clinical practices.

DETAILED DESCRIPTION:
The Baseline visit is defined as the first office visit where an eye care professional provided an in-person office biomicroscopy exam to the subject, before or during which a TOTAL30 sphere or toric contact lens prescription was released. Baseline visit data will be collected retrospectively (chart review).

The Year 1 visit is defined as the visit that occurs 1 year (-2/+6 months) since the Baseline visit during which period the subject is wearing test lenses of the same design in both eyes, and a contact lens examination is performed. Year 1 data will be collected either retrospectively or prospectively (eye exam).

ELIGIBILITY:
Key Inclusion Criteria:

* Wearers of lehfilcon A (sphere or toric) contact lenses of the same design in both eyes who have already begun use of the lens type and have purchased at least 3-month supply of lenses at the baseline timepoint;
* Best corrected spectacle visual acuity (VA) 20/25 or better at baseline;
* Healthy, non-diseased eyes;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria, as determined or known by the Investigator:

* Any ocular disease or condition that would contraindicate contact lens wear present at baseline;
* The use of systemic or ocular medications that would contraindicate contact lens wear at baseline;
* Participation in a contact lens or contact lens care product clinical trial during the period of the retrospective chart collection or during prospective study participation;
* Other protocol-specified exclusion criteria may apply.

Min Age: 7 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from clinical sites located in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity with study lenses at baseline | Baseline
  Visual acuity (VA) assessed per the investigator's standard of care with study lenses in place.
Distance visual acuity with study lenses at 1-year follow-up | Year 1
  Visual acuity (VA) assessed per the investigator's standard of care with study lenses in place.
Incidence of corneal infiltrative events | Up to Year 1
  Incidence of corneal infiltrative events occurring after the Baseline Visit will be determined retrospectively (chart review) and prospectively (eye exam).
Incidence of microbial keratitis | Up to Year 1
  Incidence of microbial keratitis occurring after the Baseline Visit will be determined retrospectively (chart review) and prospectively (eye exam).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No